CLINICAL TRIAL: NCT05860413
Title: Intermittent Fasting for the Treatment of Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Felicia Steger, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00149127
Record Dates: First submitted 2023-02-23; First posted 2023-05-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent energy restriction (IER) (Experimental): Intermittent fasting using a very-low energy diet (VLED; 550-800 kcal/d) 2-3 days per week
  Interventions: Behavioral: Intermittent energy restriction (IER)
- Time-restricted eating (TRE) (Experimental): Intermittent fasting using an 8-hour eating period.
  Interventions: Behavioral: Time Restricted Eating (TRE)

INTERVENTIONS:
Behavioral: Intermittent energy restriction (IER) — During Phase 1 (Weight Loss), participants will follow a very-low energy diet (VLED; 550-800 kcal/d) 2-3 days per week. On other days, participants do not have a specific kcal goal (non-fasting days). After Phase 1, IER participants will be instructed to follow a VLED 1-2 days per week as needed for weight maintenance.
  Arms: Intermittent energy restriction (IER)
Behavioral: Time Restricted Eating (TRE) — Participants will eat within an 8-hour period most days (at least 5 days per week). All foods and beverages containing calories will be restricted to this 8-hour period but calorie-free beverages (coffee, tea, diet soda, etc.) are allowed at any time. TRE participants will follow healthy eating guidelines for weight loss during Phase 1 but not follow a specific kcal prescription or restrict intake thereafter.
  Arms: Time-restricted eating (TRE)

SUMMARY:
To test whether a lifestyle program featuring one of two forms of intermittent fasting (IER or TRE) can feasibly and effectively improve glycemia in patients with type 2 diabetes, and potentially induce diabetes remission.

DETAILED DESCRIPTION:
Intermittent energy restriction (IER) and time-restricted eating (TRE) are two distinct forms of intermittent fasting which have yet to be compared for the treatment of type 2 diabetes. Investigators will test whether a comprehensive, intensive lifestyle program featuring each of these intermittent fasting approaches is feasible and effective for improving glycemic control in patients diagnosed with type 2 diabetes within the past 10 years. Both interventions will be delivered over one year in three phases: (1) a 12-week weight loss program featuring weekly group meetings, (2) a 12-week weight maintenance program featuring biweekly group meetings, and (3) a 6-month low-contact follow up period featuring monthly check-ins.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes in the past 10 years.
2. Age 21-65 years
3. BMI of 25 - 45 kg/m2
4. HbA1c of 6.7-9.5%, or those with A1c of <6.7% on glucose-lowering medications
5. Ability to participate in a graduated physical activity program
6. Clearance from study physician.

Exclusion Criteria:

1. Inability to attend health education meetings.
2. Weight change of >=5% in the previous 3 months.
3. Addition of new antihyperglycemic or weight-reducing medication in the previous 2 months.
4. Serious medical risk such as ongoing treatment for cancer, uncontrolled hypertension, recent cardiac event, or other medical condition presenting acute risk of participation in a lifestyle change program.
5. Untreated depression or anxiety, or increase in associated medications in the previous 3 months.
6. Current participation in another lifestyle change intervention, such as a tobacco cessation program or physical activity program.
7. Pregnancy or lactation within the previous six months
8. Weight of >450 lbs
9. Currently taking medications that may result in hypoglycemia during fasting and unwilling to stop prior to the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Retention | 52 weeks
  Feasibility of IER and TRE over one year assessed by retention (# completed / # enrolled) and attendance (# classes attended / # classes offered).
Adherence to diet protocols | Weekly from baseline to 52 weeks
  Acceptability of IER and TRE over one year as assessed by compliance to program recommendations (# weeks adhered / # study weeks).

SECONDARY OUTCOMES:
HbA1c | Change from baseline to 24 weeks
  Estimate the effects for both IER and TRE on long-term glycemic control assessed via HbA1c
Oral Glucose Tolerance Test | Change from baseline to 24 weeks
  Estimate the effects for both IER and TRE on fasting and 3 hr glucose result.
Isulin resistance | Change from baseline to 24 weeks
  Estimate the effects for both IER and TRE on insulin resistance estimated by the oral minimal model during a mixed meal tolerance test
Insulin sensitivity | Change from baseline to 24 weeks
  Estimate the effects for both IER and TRE on insulin sensitivity estimated by the oral minimal model during a mixed meal tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF